CLINICAL TRIAL: NCT05704075
Title: Clinical and Mechanistic Study of Transverse Tibial Transport in Complex Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Samuel KK Ling, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTTFootUlcers
Record Dates: First submitted 2022-10-13; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): Conventional Treatment: Dressing + Negative Pressure Wound Therapy
  Interventions: Procedure: Conventional
- TTT Group (Experimental): Dressing + Negative Pressure Wound Therapy + Transverse Tibial Transport
  Interventions: Procedure: Transverse Tibial Transport (TTT)

INTERVENTIONS:
Procedure: Transverse Tibial Transport (TTT) — Transverse tibial transport is a novel adaptation of concepts used in distraction histogenesis. The most common use of this surgical principle is in bone lengthening surgery, which is a well-established surgical procedure by applying an external fixator to the bone, creating a corticotomy, and gradually lengthening the bone at the optimal rate of 0.5mm/12hrs. The biological mechanisms of distraction histogenesis involve activating signalling pathways such as cytokines Interleukin 1 and Interleukin 6, pro-inflammatory markers TNF alpha, pro-osteogenic TGF-beta, BMPs and pro-angiogenic factors VEGF and angiopoietin . TTT utilises the concept of distraction histiogenesis, but distraction is performed in the transverse plane instead of a longitudinal distraction. In addition, the period of distraction is coupled with a corresponding compression period and ultimately results in no net change in limb length.
  Arms: TTT Group
Procedure: Conventional — Dressing + Negative Pressure Wound Therapy
  Arms: Control Group

SUMMARY:
TTT is a novel surgical technique that may potentially solve the long-standing deficit of seeking effective treatment for diabetic foot ulcers, decreasing the need for amputations and softening the socio-economic impact it brings. This trial will be the world's first prospective RCT to verify the promising clinical studies on the clinical benefit of TTT in treating diabetic foot ulcers. In addition, blood samples from this study will allow us to study the various systemic circulating soluble factors in relation to neovascularisation, immunomodulation, and stem cell mobilisation. By taking the blood and various time points, we will better understand the complex interplay between various biomarkers. This GRF will allow us to obtain tissue samples to analyse the histological cellular changes after TTT surgery. It will provide us with more insight on how TTT works, as well as potentially helping us pinpoint the important changes and timeframes related to this intervention.

The PI, Co-Is and collaborators create a strong team of clinicians and scientists with a solid clinical and basic science track record. The team has published guidelines and surgical techniques in TTT and run several training cadaveric workshops teaching the TTT surgical technique to local orthopaedic surgeons. The team has also established a rat TTT model and published on TTT immunomodulation and neovascularisation in addition to other ongoing mechanistic experiments in animals.

This prospective multi-centre randomised controlled trial may act as the foundation for launching this cost-effective TTT surgery to regulate neovascularisation, neurogenesis, immunomodulation and mobilisation of MSCs for the treatment of various chronic conditions. Regenerative medicine is a multi-million dollar industry, and the potential use of TTT can result in a range of clinical applications not limited to DFUs.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years old
* Patients with a Wagner stage 4 Foot ulcer (partial foot gangrene)
* No active wound infection as confirmed by bacterial fluorescence imaging. (the Moleculight i:X, Smith and Nephew handheld device illuminates with 405nm violet light which causes bacteria to emit characteristic endogenous fluorescence signals that are visualised in real-time on the device's screen, allowing an objective measure of adequate surgical debridement)
* Biochemically confirmed diabetes with fasting plasma glucose ≥ 7.0 mmol/L, or a random plasma glucose ≥ 11.1 mmol/L or haemoglobin A1c (HbA1c) level ≥ 6.5%
* Triaged out for angioplasty/vascular bypass by the vascular surgeon
* Triaged out of reconstructive flap surgery by the microvascular surgeon

Exclusion Criteria:

* Uncontrolled sepsis
* Contraindications for applying an external fixator device in the tibia (overlying skin conditions, surgical hardware such as tibial nails, total knee prosthesis etc.)
* Severe medical comorbidities precluding safe anaesthesia (recent myocardial infarct, limited pulmonary function etc.)
* Mental or physical disability which may impair the ability to adhere to the intervention plan, e.g. severe dementia, psychosis etc.
* Recent revascularisation procedure (<12 weeks)
* Recent medication/intervention affecting cell proliferation (e.g. chemotherapy, radiotherapy etc.), radiotherapy etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Wound Size | 0 month
  Wound size will be measured using digital photography with standardised marker dots.
Wound Size | 1 month
  Wound size will be measured using digital photography with standardised marker dots.
Wound Size | 3 month
  Wound size will be measured using digital photography with standardised marker dots.
Wound Size | 6 month
  Wound size will be measured using digital photography with standardised marker dots.
Wound Size | 12 month
  Wound size will be measured using digital photography with standardised marker dots.

SECONDARY OUTCOMES:
Foot Function | 0 month
  Foot function will be objectively measured using our validated Chinese Foot and Ankle Outcome Score or the original English version.
Foot Function | 1 month
  Foot function will be objectively measured using our validated Chinese Foot and Ankle Outcome Score or the original English version.
Foot Function | 3 month
  Foot function will be objectively measured using our validated Chinese Foot and Ankle Outcome Score or the original English version.
Foot Function | 6 month
  Foot function will be objectively measured using our validated Chinese Foot and Ankle Outcome Score or the original English version.
Foot Function | 12 month
  Foot function will be objectively measured using our validated Chinese Foot and Ankle Outcome Score or the original English version.
Incidence of Amputation | Up to 52 weeks
  Incidence of Amputation
Ankle Brachial Pressure Index | 0 month
  The ankle brachial pressure index (API) is a clinical measurement of peripheral vascular perfusion.
Ankle Brachial Pressure Index | 1 month
  The ankle brachial pressure index (API) is a clinical measurement of peripheral vascular perfusion.
Ankle Brachial Pressure Index | 3 month
  The ankle brachial pressure index (API) is a clinical measurement of peripheral vascular perfusion.
Ankle Brachial Pressure Index | 6 month
  The ankle brachial pressure index (API) is a clinical measurement of peripheral vascular perfusion.
Ankle Brachial Pressure Index | 12 month
  The ankle brachial pressure index (API) is a clinical measurement of peripheral vascular perfusion.
ELISA of angiogenic factors | 0 month
  10ml peripheral blood samples will be collected at multiple time points and human serum vascular endothelial growth factor (VEGF), basic fibroblast growth factor (bFGF), epidermal growth factor (EGF), and platelet-derived growth factor (PDGF) will be analysed with an ELISA kit was processed according to its protocol.
ELISA of angiogenic factors | 1 month
  10ml peripheral blood samples will be collected at multiple time points and human serum vascular endothelial growth factor (VEGF), basic fibroblast growth factor (bFGF), epidermal growth factor (EGF), and platelet-derived growth factor (PDGF) will be analysed with an ELISA kit was processed according to its protocol.
ELISA of angiogenic factors | 3 month
  10ml peripheral blood samples will be collected at multiple time points and human serum vascular endothelial growth factor (VEGF), basic fibroblast growth factor (bFGF), epidermal growth factor (EGF), and platelet-derived growth factor (PDGF) will be analysed with an ELISA kit was processed according to its protocol.
ELISA of angiogenic factors | 6 month
  10ml peripheral blood samples will be collected at multiple time points and human serum vascular endothelial growth factor (VEGF), basic fibroblast growth factor (bFGF), epidermal growth factor (EGF), and platelet-derived growth factor (PDGF) will be analysed with an ELISA kit was processed according to its protocol.
ELISA of angiogenic factors | 12 month
  10ml peripheral blood samples will be collected at multiple time points and human serum vascular endothelial growth factor (VEGF), basic fibroblast growth factor (bFGF), epidermal growth factor (EGF), and platelet-derived growth factor (PDGF) will be analysed with an ELISA kit was processed according to its protocol.
Immunostaining of angiogenic markers | 0 month
  3mm punch biopsy (RazorMed) will be obtained from the wound edge at multiple timepoints. The samples will be processed for paraffin embedding and 7μm serial thin sections will be cut. Markers for angiogenesis (CD31, alpha-SMA) and cell proliferation (Ki-67) antibodies will be used for immunostaining on the paraffin section according to the previously published protocol. The positively stained cell numbers in the DFU zone in each patient will be quantified using imaging software according to published protocol. The paired T test will be adopted to compare the difference of MSCs proportion, angiogenesis, and cell proliferation in each patient by SPSS 18.0 software for windows (SPSS, Chicago, IL, USA). Nonparametric test will be used for comparison of mean values with p<0.05 considered as statistically significant.
Immunostaining of angiogenic markers | 1 month
  3mm punch biopsy (RazorMed) will be obtained from the wound edge at multiple timepoints. The samples will be processed for paraffin embedding and 7μm serial thin sections will be cut. Markers for angiogenesis (CD31, alpha-SMA) and cell proliferation (Ki-67) antibodies will be used for immunostaining on the paraffin section according to the previously published protocol. The positively stained cell numbers in the DFU zone in each patient will be quantified using imaging software according to published protocol. The paired T test will be adopted to compare the difference of MSCs proportion, angiogenesis, and cell proliferation in each patient by SPSS 18.0 software for windows (SPSS, Chicago, IL, USA). Nonparametric test will be used for comparison of mean values with p<0.05 considered as statistically significant.
Immunostaining of angiogenic markers | 3 month
  3mm punch biopsy (RazorMed) will be obtained from the wound edge at multiple timepoints. The samples will be processed for paraffin embedding and 7μm serial thin sections will be cut. Markers for angiogenesis (CD31, alpha-SMA) and cell proliferation (Ki-67) antibodies will be used for immunostaining on the paraffin section according to the previously published protocol. The positively stained cell numbers in the DFU zone in each patient will be quantified using imaging software according to published protocol. The paired T test will be adopted to compare the difference of MSCs proportion, angiogenesis, and cell proliferation in each patient by SPSS 18.0 software for windows (SPSS, Chicago, IL, USA). Nonparametric test will be used for comparison of mean values with p<0.05 considered as statistically significant.
Immunostaining of angiogenic markers | 6 month
  3mm punch biopsy (RazorMed) will be obtained from the wound edge at multiple timepoints. The samples will be processed for paraffin embedding and 7μm serial thin sections will be cut. Markers for angiogenesis (CD31, alpha-SMA) and cell proliferation (Ki-67) antibodies will be used for immunostaining on the paraffin section according to the previously published protocol. The positively stained cell numbers in the DFU zone in each patient will be quantified using imaging software according to published protocol. The paired T test will be adopted to compare the difference of MSCs proportion, angiogenesis, and cell proliferation in each patient by SPSS 18.0 software for windows (SPSS, Chicago, IL, USA). Nonparametric test will be used for comparison of mean values with p<0.05 considered as statistically significant.
Immunostaining of angiogenic markers | 12 month
  3mm punch biopsy (RazorMed) will be obtained from the wound edge at multiple timepoints. The samples will be processed for paraffin embedding and 7μm serial thin sections will be cut. Markers for angiogenesis (CD31, alpha-SMA) and cell proliferation (Ki-67) antibodies will be used for immunostaining on the paraffin section according to the previously published protocol. The positively stained cell numbers in the DFU zone in each patient will be quantified using imaging software according to published protocol. The paired T test will be adopted to compare the difference of MSCs proportion, angiogenesis, and cell proliferation in each patient by SPSS 18.0 software for windows (SPSS, Chicago, IL, USA). Nonparametric test will be used for comparison of mean values with p<0.05 considered as statistically significant.
Semmes Weinstein monofilament test | 0 month
  a monofilament sized 0.57, with a buckling force of 10gm, is the clinically accepted cutoff for the presence or absence of protective sensation. Measurements will be standardised to 3 sites; the 1st metatarsal, 3rd metatarsal and 5th metatarsal.
Semmes Weinstein monofilament test | 1 month
  a monofilament sized 0.57, with a buckling force of 10gm, is the clinically accepted cutoff for the presence or absence of protective sensation. Measurements will be standardised to 3 sites; the 1st metatarsal, 3rd metatarsal and 5th metatarsal.
Semmes Weinstein monofilament test | 3 month
  a monofilament sized 0.57, with a buckling force of 10gm, is the clinically accepted cutoff for the presence or absence of protective sensation. Measurements will be standardised to 3 sites; the 1st metatarsal, 3rd metatarsal and 5th metatarsal.
Semmes Weinstein monofilament test | 6 month
  a monofilament sized 0.57, with a buckling force of 10gm, is the clinically accepted cutoff for the presence or absence of protective sensation. Measurements will be standardised to 3 sites; the 1st metatarsal, 3rd metatarsal and 5th metatarsal.
Semmes Weinstein monofilament test | 12 month
  a monofilament sized 0.57, with a buckling force of 10gm, is the clinically accepted cutoff for the presence or absence of protective sensation. Measurements will be standardised to 3 sites; the 1st metatarsal, 3rd metatarsal and 5th metatarsal.
Section of neurogenic markers | 0 month
  3mm punch biopsy (RazorMed) will be obtained from the wound edge at multiple timepoints. The samples will be processed for paraffin embedding and 7μm serial thin sections will be cut. The samples will be dewaxed and rehydrated. After antigen recovery (by Citrate Antigen Retrieval solution, ~30min, 65℃) and Permeabilization (by Triton™ X-100), markers for axon (beta-tubulin 3) (38) will be incubated overnight and corresponding secondary antibody will be incubated for 1 hours. The positively stained area in the DFU zone in each patient will be quantified using imaging software according to published protocol. The paired T test will be adopted to compare the difference of axon area in each patient by SPSS 18.0 software for windows (SPSS, Chicago, IL, USA). Nonparametric test will be used for comparison of mean values with p<0.05 considered as statistically significant.
Section of neurogenic markers | 1 month
  3mm punch biopsy (RazorMed) will be obtained from the wound edge at multiple timepoints. The samples will be processed for paraffin embedding and 7μm serial thin sections will be cut. The samples will be dewaxed and rehydrated. After antigen recovery (by Citrate Antigen Retrieval solution, ~30min, 65℃) and Permeabilization (by Triton™ X-100), markers for axon (beta-tubulin 3) (38) will be incubated overnight and corresponding secondary antibody will be incubated for 1 hours. The positively stained area in the DFU zone in each patient will be quantified using imaging software according to published protocol. The paired T test will be adopted to compare the difference of axon area in each patient by SPSS 18.0 software for windows (SPSS, Chicago, IL, USA). Nonparametric test will be used for comparison of mean values with p<0.05 considered as statistically significant.
Section of neurogenic markers | 3 month
  3mm punch biopsy (RazorMed) will be obtained from the wound edge at multiple timepoints. The samples will be processed for paraffin embedding and 7μm serial thin sections will be cut. The samples will be dewaxed and rehydrated. After antigen recovery (by Citrate Antigen Retrieval solution, ~30min, 65℃) and Permeabilization (by Triton™ X-100), markers for axon (beta-tubulin 3) (38) will be incubated overnight and corresponding secondary antibody will be incubated for 1 hours. The positively stained area in the DFU zone in each patient will be quantified using imaging software according to published protocol. The paired T test will be adopted to compare the difference of axon area in each patient by SPSS 18.0 software for windows (SPSS, Chicago, IL, USA). Nonparametric test will be used for comparison of mean values with p<0.05 considered as statistically significant.
Section of neurogenic markers | 6 month
  3mm punch biopsy (RazorMed) will be obtained from the wound edge at multiple timepoints. The samples will be processed for paraffin embedding and 7μm serial thin sections will be cut. The samples will be dewaxed and rehydrated. After antigen recovery (by Citrate Antigen Retrieval solution, ~30min, 65℃) and Permeabilization (by Triton™ X-100), markers for axon (beta-tubulin 3) (38) will be incubated overnight and corresponding secondary antibody will be incubated for 1 hours. The positively stained area in the DFU zone in each patient will be quantified using imaging software according to published protocol. The paired T test will be adopted to compare the difference of axon area in each patient by SPSS 18.0 software for windows (SPSS, Chicago, IL, USA). Nonparametric test will be used for comparison of mean values with p<0.05 considered as statistically significant.
Section of neurogenic markers | 12 month
  3mm punch biopsy (RazorMed) will be obtained from the wound edge at multiple timepoints. The samples will be processed for paraffin embedding and 7μm serial thin sections will be cut. The samples will be dewaxed and rehydrated. After antigen recovery (by Citrate Antigen Retrieval solution, ~30min, 65℃) and Permeabilization (by Triton™ X-100), markers for axon (beta-tubulin 3) (38) will be incubated overnight and corresponding secondary antibody will be incubated for 1 hours. The positively stained area in the DFU zone in each patient will be quantified using imaging software according to published protocol. The paired T test will be adopted to compare the difference of axon area in each patient by SPSS 18.0 software for windows (SPSS, Chicago, IL, USA). Nonparametric test will be used for comparison of mean values with p<0.05 considered as statistically significant.
Inflammatory cell flow cytometry | 0 month
  10ml of peripheral blood will be obtained. Mononuclear cells will be collected by isolation of Ficoll-Paque density gradient centrifugation. The populations of classical and non-classical monocytes will be analyzed by flow cytometry and identified from proportions of CD172a+ and CD43+ cells.
Inflammatory cell flow cytometry | 1 month
  10ml of peripheral blood will be obtained. Mononuclear cells will be collected by isolation of Ficoll-Paque density gradient centrifugation. The populations of classical and non-classical monocytes will be analyzed by flow cytometry and identified from proportions of CD172a+ and CD43+ cells.
Inflammatory cell flow cytometry | 3 month
  10ml of peripheral blood will be obtained. Mononuclear cells will be collected by isolation of Ficoll-Paque density gradient centrifugation. The populations of classical and non-classical monocytes will be analyzed by flow cytometry and identified from proportions of CD172a+ and CD43+ cells.
Inflammatory cell flow cytometry | 6 month
  10ml of peripheral blood will be obtained. Mononuclear cells will be collected by isolation of Ficoll-Paque density gradient centrifugation. The populations of classical and non-classical monocytes will be analyzed by flow cytometry and identified from proportions of CD172a+ and CD43+ cells.
Inflammatory cell flow cytometry | 12 month
  10ml of peripheral blood will be obtained. Mononuclear cells will be collected by isolation of Ficoll-Paque density gradient centrifugation. The populations of classical and non-classical monocytes will be analyzed by flow cytometry and identified from proportions of CD172a+ and CD43+ cells.
Macrophage Immunofluorescence staining | 0 month
  A 3mm punch biopsy (RazorMed) will be obtained and prepared for paraffin sections. The populations and localisations of both monocytes (classical and non-classical phenotypes) and macrophages (M1 and M2 phenotype) in the skin wound site will be determined by immunofluorescence staining with specific antibodies to CD68 (general marker for macrophage), anti-iNOS (M1 macrophage), CD206 (M2 macrophage) [32] CD172a (general marker for monocyte) and CD43 (non-classical monocyte specific marker).
Macrophage Immunofluorescence staining | 1 month
  A 3mm punch biopsy (RazorMed) will be obtained and prepared for paraffin sections. The populations and localisations of both monocytes (classical and non-classical phenotypes) and macrophages (M1 and M2 phenotype) in the skin wound site will be determined by immunofluorescence staining with specific antibodies to CD68 (general marker for macrophage), anti-iNOS (M1 macrophage), CD206 (M2 macrophage) [32] CD172a (general marker for monocyte) and CD43 (non-classical monocyte specific marker).
Macrophage Immunofluorescence staining | 3 month
  A 3mm punch biopsy (RazorMed) will be obtained and prepared for paraffin sections. The populations and localisations of both monocytes (classical and non-classical phenotypes) and macrophages (M1 and M2 phenotype) in the skin wound site will be determined by immunofluorescence staining with specific antibodies to CD68 (general marker for macrophage), anti-iNOS (M1 macrophage), CD206 (M2 macrophage) [32] CD172a (general marker for monocyte) and CD43 (non-classical monocyte specific marker).
Macrophage Immunofluorescence staining | 6 month
  A 3mm punch biopsy (RazorMed) will be obtained and prepared for paraffin sections. The populations and localisations of both monocytes (classical and non-classical phenotypes) and macrophages (M1 and M2 phenotype) in the skin wound site will be determined by immunofluorescence staining with specific antibodies to CD68 (general marker for macrophage), anti-iNOS (M1 macrophage), CD206 (M2 macrophage) [32] CD172a (general marker for monocyte) and CD43 (non-classical monocyte specific marker).
Macrophage Immunofluorescence staining | 12 month
  A 3mm punch biopsy (RazorMed) will be obtained and prepared for paraffin sections. The populations and localisations of both monocytes (classical and non-classical phenotypes) and macrophages (M1 and M2 phenotype) in the skin wound site will be determined by immunofluorescence staining with specific antibodies to CD68 (general marker for macrophage), anti-iNOS (M1 macrophage), CD206 (M2 macrophage) [32] CD172a (general marker for monocyte) and CD43 (non-classical monocyte specific marker).
Identification of regulatory cytokines for peripheral blood mesenchymal stem cells (PB-MSCs) mobilization | 0 month
  10ml of peripheral blood will be collected at multiple timepoints. Each peripheral blood samples will be collected using tubes containing K2-EDTA. Blood samples will be centrifuged at 1800g for 6 min at 4 °C to get plasma and apportioned into 1 mL aliquots and stored at -80 °C. Differential protein expression will be determined by 8-plex isobaric tags for relative and absolute quantitation (iTRAQ)-based quantitative proteomics analysis.
Identification of regulatory cytokines for peripheral blood mesenchymal stem cells (PB-MSCs) mobilization | 1 month
  10ml of peripheral blood will be collected at multiple timepoints. Each peripheral blood samples will be collected using tubes containing K2-EDTA. Blood samples will be centrifuged at 1800g for 6 min at 4 °C to get plasma and apportioned into 1 mL aliquots and stored at -80 °C. Differential protein expression will be determined by 8-plex isobaric tags for relative and absolute quantitation (iTRAQ)-based quantitative proteomics analysis.
Identification of regulatory cytokines for peripheral blood mesenchymal stem cells (PB-MSCs) mobilization | 3 month
  10ml of peripheral blood will be collected at multiple timepoints. Each peripheral blood samples will be collected using tubes containing K2-EDTA. Blood samples will be centrifuged at 1800g for 6 min at 4 °C to get plasma and apportioned into 1 mL aliquots and stored at -80 °C. Differential protein expression will be determined by 8-plex isobaric tags for relative and absolute quantitation (iTRAQ)-based quantitative proteomics analysis.
Identification of regulatory cytokines for peripheral blood mesenchymal stem cells (PB-MSCs) mobilization | 6 month
  10ml of peripheral blood will be collected at multiple timepoints. Each peripheral blood samples will be collected using tubes containing K2-EDTA. Blood samples will be centrifuged at 1800g for 6 min at 4 °C to get plasma and apportioned into 1 mL aliquots and stored at -80 °C. Differential protein expression will be determined by 8-plex isobaric tags for relative and absolute quantitation (iTRAQ)-based quantitative proteomics analysis.
Identification of regulatory cytokines for peripheral blood mesenchymal stem cells (PB-MSCs) mobilization | 12 month
  10ml of peripheral blood will be collected at multiple timepoints. Each peripheral blood samples will be collected using tubes containing K2-EDTA. Blood samples will be centrifuged at 1800g for 6 min at 4 °C to get plasma and apportioned into 1 mL aliquots and stored at -80 °C. Differential protein expression will be determined by 8-plex isobaric tags for relative and absolute quantitation (iTRAQ)-based quantitative proteomics analysis.